CLINICAL TRIAL: NCT02306759
Title: Ketamine For Acute Treatment of Pain in Emergency Department
Acronym: KETAFAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Brooklyn Hospital Center (Other)
Responsible Party: Principal Investigator, Billy Sin, Emergency Medicine Clinical Pharmacy Educator, The Brooklyn Hospital Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 669443-1
Record Dates: First submitted 2014-11-25; First posted 2014-12-03 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Pain
Keywords: analgesia; ketamine; pain
MeSH Terms: conditions — Pain; Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Ketamine 0.3mg/kg intravenous piggyback (IVPB) in 50ml NS over 15 minutes Morphine 0.1mg/kg intravenous push (IVP) PRN at designated intervals
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Normal saline 50ml intravenous piggyback (IVPB) over 15 minutes Morphine 0.1mg/kg intravenous push (IVP) PRN at designated intervals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine 0.3mg/kg in 50ml normal saline, administered over 15 minutes
  Arms: Treatment
Drug: Placebo — Normal saline 50ml, administered over 15 minutes
  Arms: Placebo

SUMMARY:
The aim of the study is to compare the safety & efficacy of low dose ketamine and morphine versus morphine alone for acute generalized pain in the Emergency Department (ED). The investigators are also interested to investigate whether low-dose ketamine is a safe and effective alternative option to opioids for the acute treatment of pain in the Emergency Department.

The agents that are available in the department includes acetaminophen, non-steroidal anti-inflammatory (NSAIDS) and opioids. In most cases, acetaminophen and NSAIDS are not adequate to manage acute pain crisis. There is also heightening concerns for increased opioid use or abuse by patients. Since the HCAPHS survey includes various questions which inquires about patient perception of pain management in the department, the investigators are interested in investigating the safety and efficacy of low-dose ketamine to as an alternative method to opioids for the acute management of pain. There has been limited, mostly observational pilot studies, published in the literature. Limited data in the literature have reported the incidence of nausea and vomiting ranged from 3-13%. All published literature administered low-dose ketamine as an intravenous push. To the best of our knowledge our study would be the first study to administer low-dose ketamine as a short bolus infusion to mitigate the incidence of nausea and vomiting. The investigators believe our study would provide important scientific data to fill the theoretical gap that low-dose ketamine at 0.3mg/kg/dose may be a safe and effective agent for acute pain management in an ED that is located in the center of a densely populated urban area.

DETAILED DESCRIPTION:
The aim of the study is to compare the safety & efficacy of low dose ketamine and morphine versus morphine alone for acute generalized pain in the Emergency Department (ED). The is a randomized double blind placebo controlled trial to investigate the effects of low dose ketamine and morphine versus placebo and morphine for the management of acute pain in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older presenting with acute generalized pain
* Describes pain to be greater than or equal to 3 on the Visual Analogue Scale (VAS)
* Provides informed consent

Exclusion Criteria:

* Patients who are admitted to the hospital
* Severe hypertension(≥180/100)
* Presence of or suspected for traumatic head injury with or without loss of consciousness
* Presence of or suspected for myocardial ischemia
* Presence of or suspected alcohol intoxication
* Hemodynamic instability
* History of schizophrenia
* History of Sickle cell crisis / presenting with acute sickle cell crisis
* History of or suspected recreational substance abuse
* History of or suspected diagnosis of headache or migraine
* History of or suspected diagnosis increase in intracranial/intraocular pressure
* Known or suspected pregnancy
* Allergy to ketamine or morphine
* Administration of opioids in previous 4 hours
* Patients with language barriers or in altered mental status who are unable to describe pain
* Patients weighing over 166kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Billy Sin, Pharm.D., Principal Investigator — The Brooklyn Hospital Center
Locations (1):
- The Brooklyn Hospital Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Gurnani A, Sharma PK, Rautela RS, Bhattacharya A. Analgesia for acute musculoskeletal trauma: low-dose subcutaneous infusion of ketamine. Anaesth Intensive Care. 1996 Feb;24(1):32-6. doi: 10.1177/0310057X9602400106. PMID 8669651
- [Background] Yeaman F, Oakley E, Meek R, Graudins A. Sub-dissociative dose intranasal ketamine for limb injury pain in children in the emergency department: a pilot study. Emerg Med Australas. 2013 Apr;25(2):161-7. doi: 10.1111/1742-6723.12059. Epub 2013 Mar 20. PMID 23560967
- [Background] Yeaman F, Meek R, Egerton-Warburton D, Rosengarten P, Graudins A. Sub-dissociative-dose intranasal ketamine for moderate to severe pain in adult emergency department patients. Emerg Med Australas. 2014 Jun;26(3):237-42. doi: 10.1111/1742-6723.12173. Epub 2014 Apr 8. PMID 24712757
- [Background] Ahern TL, Herring AA, Stone MB, Frazee BW. Effective analgesia with low-dose ketamine and reduced dose hydromorphone in ED patients with severe pain. Am J Emerg Med. 2013 May;31(5):847-51. doi: 10.1016/j.ajem.2013.02.008. Epub 2013 Apr 18. PMID 23602757
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center, prospective, randomized, double-blind, placebo-controlled trial comparing the use of SDDK versus placebo as an adjunct therapy for moderate to severe acute pain in the ED. The study was conducted in a community teaching hospital with a level-2 trauma ED where more than 77,000 patients are treated annually.
Groups:
- Treatment: Ketamine 0.3mg/kg IVPB in 50ml NS over 15 minutes Morphine 0.1mg/kg IVP PRN at designated intervals
  Ketamine: Ketamine 0.3mg/kg in 50ml normal saline, administered over 15 minutes
- Placebo: Normal saline 50ml IVPB over 15 minutes Morphine 0.1mg/kg IVP PRN at designated intervals
  Placebo: Normal saline 50ml, administered over 15 minutes
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (16) | 48 (17) | 44 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Pain as Described by Numeric Rating Scale (NRS) [Minimum:0, Maximum 10] at 15 Minutes
Description: Change from Baseline of Pain as described by Numeric Rating Scale (NRS) [minimum:0, maximum 10] at 15 minutes. Lower values indicate worst outcomes while higher values indicate better outcomes.
Time Frame: 15 minutes after administration of study intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Treatment: Ketamine 0.3mg/kg intravenous piggyback (IVPB) in 50ml NS over 15 minutes
  Morphine 0.1mg/kg intravenous push (IVP) PRN at designated intervals
  Ketamine: Ketamine 0.3mg/kg in 50ml normal saline, administered over 15 minutes
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 3.5 [1.0 to 7.3] | 6.0 [4.0 to 9.0]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Incidence or number of participants with adverse events.
Time Frame: during the study period
Population: Nausea was reported in three patients who received placebo and one patient who received ketamine. Dreams was reported in 1 patient who received placebo and one patient who received ketamine.
Measure: Number; unit: participants
Groups:
- Treatment: Ketamine 0.3mg/kg IVPB in 50ml NS over 15 minutes Morphine 0.1mg/kg IVP PRN at designated intervals
- Placebo: Normal saline 50ml IVPB over 15 minutes Morphine 0.1mg/kg IVP PRN at designated intervals
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 30 | 30
participants | 2 | 4

3. Secondary Outcome: Patient Satisfaction of Pain Control Based on a Likert Scale
Description: Patient satisfaction of pain control based on a Likert Scale at the end of study completion, an average of 90 minutes. Scores reported out of scale of 10, 10 being most satisfied and 1 being least satisfied.
Time Frame: At the end of study period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 8.57 (2.1) | 6.05 (2.6)

4. Secondary Outcome: Mean Consumption of Rescue Analgesia
Time Frame: at designated intervals during study period (0, 15, 30, 45, 60, 75, 90, 105, 120 minutes)
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 30 | 30
milligrams
  T5 | 0 (0) | 0 (0)
  T15 | 0.23 (1.3) | 0.14 (0.74)
  T30 | 0.37 (1.45) | 0.28 (1.03)
  T45 | 0.07 (0.37) | 0 (0)
  T60 | 0 (0) | 0.22 (1.15)
  T75 | 0 (0) | 0 (0)
  T90 | 0.48 (1.66) | 0 (0)
  T105 | 0.55 (1.87) | 0.42 (1.26)
  T120 | 0 (0) | 0.42 (1.7)

5. Secondary Outcome: ED Length of Stay (Minutes)
Description: ED Length of stay (minutes) throughout study period
Time Frame: throughout study completion
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 30 | 30
minutes | 267 (191) | 292 (203)

ADVERSE EVENTS:
Arm/Group | Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30) | Placebo (N=30)
Dreams (Nervous system disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) — Nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes